CLINICAL TRIAL: NCT00238758
Title: A Randomised, Double-Blind, Placebo Controlled Trial of Omega-3 Polyunsaturated Fatty Acids as a Monotherapy for Major Depression
Brief Title: A Study of Omega-3 as a Treatment for Major Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Your Health Inc. (Other); Sphere Healthcare (Industry); Ocean Nutrition (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05157
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Major Depression; Dysthymia
Keywords: Mood Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Mood Disorders | interventions — Docosahexaenoic Acids

INTERVENTIONS:
Drug: Omega-3 Polyunsaturated Fatty Acids

SUMMARY:
The purpose of this study is to determine whether omega-3 polyunsaturated fatty acids are effective as a monotherapy for depression.

DETAILED DESCRIPTION:
The study will be a 6 week, parallel-group, double-blind randomized controlled trial of the efficacy of Omega-3 as a monotherapy for depression. People aged 21-65 who have major depression but are not currently on an antidepressant or planning to take an antidepressant in the next 14 weeks will be recruited. Participants will be randomly allocated to receive Omega-3 (fish oil) or placebo (paraffin oil) for 6 weeks. Participants will be followed up weekly and will be asked to rate their mood daily for the 6 week study period. Blood samples will be taken pre and post treatment to measure change in omega-3 levels. At the end of 6 weeks all participants will receive a further 8 weeks supply of omega-3.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM IV criteria for non-psychotic major depression lasting at least 6 weeks or dysthymia.
* Must be under the care of a mental health practitioner.
* Must be able to give informed consent.
* Must be able to attend the Black Dog Institute.

Exclusion Criteria:

* Unsuccessful treatment with more than 2 antidepressant medications (at therapeutically adequate doses and duration.
* History of psychosis or mania/hypomania or personality disorder.
* Non-English speaking or otherwise unable to provide historical information.
* Having taken Omega-3 dietary supplements in the last 3 months.
* Taking antidepressant medication for depression.
* History of allergy to n-3 PUFA supplements, finfish or shellfish.
* Pregnancy, breast feeding or planning to become pregnant during course of study.
* Post-natal depression.
* Current drug or alcohol abuse or dependence or history of abuse or dependence over the last 12 months.
* Unstable thyroid function
* Hepatic or renal impairment or other medical conditions that may interfere with the absorption and metabolism of omega-3 polyunsaturated fatty acids.
* Coagulopathy or anticoagulant treatment.
* Patients who, in the investigator's judgment pose a current serious suicidal or other safety risk, or patients who are not likely to be able to comply with the study protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2005-10

PRIMARY OUTCOMES:
Change from pretreatment score on Depression Rating Scale at 6 weeks.

SECONDARY OUTCOMES:
Weekly measure of depressive symptoms
Weekly measure of anxiety symptoms
Weekly measure of functional status

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Rees, BSc MBBS, Principal Investigator — Senior Research Fellow and Consultant Psychiatrist, School of Psychiatry, UNSW & Black Dog Institute; Gordon B Parker, Dsc MD PhD, Study Director — Professor, School of Psychiatry UNSW and Executive Director, Black Dog Institute
Locations (1):
- The University of New South Wales/ Black Dog Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Rees AM, Austin MP, Parker G. Role of omega-3 fatty acids as a treatment for depression in the perinatal period. Aust N Z J Psychiatry. 2005 Apr;39(4):274-80. doi: 10.1080/j.1440-1614.2005.01565.x. PMID 15777365
- [Background] Parker G, Gibson NA, Brotchie H, Heruc G, Rees AM, Hadzi-Pavlovic D. Omega-3 fatty acids and mood disorders. Am J Psychiatry. 2006 Jun;163(6):969-78. doi: 10.1176/ajp.2006.163.6.969. PMID 16741195
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au
- See also: University of NSW, school of psychiatry website — http://psych.med.unsw.edu.au